CLINICAL TRIAL: NCT00114998
Title: CV Disease in Adolescents With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Tom Kimball, Professor of Pediatrics, Children's Hospital Medical Center, Cincinnati
Other Study IDs: 1294; R01HL076269 (NIH)
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Heart Diseases; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To study cardiac and vascular structure and function in a population of adolescents with type 2 diabetes mellitus (T2DM) compared to a similar group with obesity alone and a similar non-obese group.

DETAILED DESCRIPTION:
BACKGROUND:

The prevalence of type 2 diabetes mellitus has increased dramatically in adolescents. This appears to be a direct result of the increase in prevalence and severity of obesity in the pediatric population. In adults with type 2 diabetes, it is well known that the risk for cardiovascular disease (CVD) is quite high. This has led to current clinical recommendation that adults with diabetes be considered equivalent in risk to those adults who already have existing coronary artery disease. It is not known if adolescents with type 2 diabetes have an equivalent high level of risk of CVD as the adult population. If they do then it would be expected that they would develop clinical CVD in their late 20's or 30's. This would have important clinical implications and would suggest the need for very aggressive management of CVD risk factors and diabetes.

DESIGN NARRATIVE:

The study is a cross-sectional evaluation of cardiac and vascular structure and function in a population of adolescents with type 2 diabetes compared to a group with similar age, sex, race and BMI with obesity alone and a non obese group with similar age, sex and race. 300 subjects with type 2 diabetes, 300 subjects with obesity and 300 non obese subjects will be studied. Assessment of CVD development will be accomplished using novel non invasive imaging methods for subclinical atherosclerosis including echocardiographic measurement of cardiac structure and function, ultrasound evaluation of carotid intimal medial thickness, and evaluation of endothelial function by brachial artery reactivity. The primary hypothesis is that adolescents with type 2 diabetes will have greater abnormality in cardiac and vascular structure and function compared to controls with obesity. Subjects with obesity alone will have greater abnormality in cardiac and vascular structure and function compared to controls who are not obese. Correlates of cardiac and vascular abnormalities including markers of inflammation, adiponectin, diet and physical activity will also be evaluated.

ELIGIBILITY:
An estimated 300 subjects, ages 10 to 23, with type 2 diabetes, 300 subjects with obesity and 300 non-obese subjects will be studied.

Inclusion Criteria:

* Diabetes, type 2
* Obese

Exclusion Criteria:

* Diabetes, type 1

Ages: 10 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Three groups of adolescents:
  1. Lean controls
  2. Obese controls (without diabetes)
  3. Obese with diabetes
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2005-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Kimball, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States